CLINICAL TRIAL: NCT00696917
Title: Safety and Immunogenicity of 3 Lots of GSK Biologicals' Novel Adjuvanted Hepatitis B Vaccine, Administered According to a 2 Dose Schedule, and Engerix™-B Administered According to a 3 Dose Schedule to Healthy Volunteers ≥ 15 Years of Age
Brief Title: Safety and Immunogenicity of 3 Lots of GSK Biologicals' HBV-MPL Vaccine and Engerix™-B in Healthy Volunteers ≥ 15y
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Isabelle Harpigny, GSK
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 208129/031
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2008-06-13 (Estimated); Status verified 2008-06

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Adjuvanted Hepatitis B vaccine; Recombinant Hepatitis B vaccine
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- Group A (Active Comparator): Three doses according to 0, 1, 6-month schedule
  Interventions: Biological: Engerix™-B
- Group B (Experimental): Two doses according to 0, 6-month schedule, with a placebo injection at Month 1
  Interventions: Biological: HBV-MPL vaccine 208129
- Group C (Experimental): Two doses according to 0, 6-month schedule, with a placebo injection at Month 1
  Interventions: Biological: HBV-MPL vaccine 208129
- Group D (Experimental): Two doses according to 0, 6-month schedule, with a placebo injection at Month 1
  Interventions: Biological: HBV-MPL vaccine 208129

INTERVENTIONS:
Biological: HBV-MPL vaccine 208129 — 2-dose intramuscular injection 3 different vaccine lots
  Arms: Group B; Group C; Group D
Biological: Engerix™-B — 3-dose intramuscular injection
  Arms: Group A

SUMMARY:
This study was conducted to evaluate the lot-to-lot consistency of three lots of HBV-MPL vaccine and to compare their safety and immunogenicity with that of Engerix™-B.

DETAILED DESCRIPTION:
At the time of conduct of this study, the sponsor GlaxoSmithKline was known by its former name SmithKline Beecham

ELIGIBILITY:
Inclusion Criteria:

* A male or female aged ≥ 15 years at the time of the first vaccination. In Centre 103 (Germany) and Centre 1 (Netherlands), only subjects ≥ 18 years will be enrolled.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Written informed consent obtained from the subject and/or from the parent or guardian of the subject.
* If the subject was a female, she was of non-childbearing potential, if of childbearing potential, she was abstinent or used adequate contraceptive precautions for one month prior to enrollment and up to two months after the last vaccination

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine (s) during the study period or within 30 days preceding the first dose of study vaccine.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before each dose of vaccine and ending 30 days after.
* Previous vaccination against hepatitis B.
* History of non-response to previous hepatitis B vaccination.
* Known exposure to hepatitis B within the past 6 weeks.
* History of hepatitis B infection.
* Confirmed human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute disease at the time of enrollment.
* Hepatomegaly, right upper quadrant abdominal pain or tenderness.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration/ administration during the study period.
* Pregnant or lactating female

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1303 (Actual)
Dates: Start 1999-04; Primary Completion 2000-02 (Actual)

PRIMARY OUTCOMES:
Occurrence, intensity and causal relationship of any (solicited/unsolicited adverse event) general symptoms | Full course of vaccination
Incidence of serious adverse events | Study period
Anti-HBs antibody concentrations | At Month 7

SECONDARY OUTCOMES:
Occurrence and intensity of solicited local signs and symptoms | 4-day after vaccination
Occurrence, intensity and relationship to vaccination of solicited general signs and symptoms | 4-day after vaccination
Occurrence, intensity and relationship to vaccination of unsolicited signs and symptoms | 30 days after vaccination
Occurrence and relationship to vaccination of SAEs | During the study period
Anti-HBs antibody concentrations | At Months 1, 2, 6 and 7

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- GSK Clinical Trials Call Center, Parkville, Victoria, Australia
- GSK Clinical Trials Call Center, Hradec Kralové, Czechia
- GSK Clinical Trials Call Center, München, Germany
- GSK Clinical Trials Call Center, Bari, Italy
- GSK Clinical Trials Call Center, Utrecht, Netherlands
- GSK Clinical Trials Call Center, Lausanne, Switzerland
- GSK Clinical Trials Call Center, London, United Kingdom